CLINICAL TRIAL: NCT07001410
Title: Geriatrics in the Intensive Care Unit. An Observational Clinical Trial
Brief Title: Geriatrics in the Intensive Care Unit
Acronym: GICU
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, MD, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2025_01_UCI_GERIATR
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Geriatrics
Keywords: Aged; Frail Older Adults; Intensive Care Units; Critical Illness; Colombia
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Younger adults: Critically ill patients, younger adults (<65 years)
  Interventions: Other: Age group
- Elders: Critically ill old patients (aged 65 to 79 years)
  Interventions: Other: Age group
- Octogenarians: Very old critically ill patients (80 years old or more)
  Interventions: Other: Age group

INTERVENTIONS:
Other: Age group — Observation of the outcomes by age groups.

SUMMARY:
Life expectancy is longer in populations of medium- and high-income countries. Older adults are an increasingly large population in intensive care units (ICUs). There are limited publications about the epidemiology, benefits, expenditure, and outcomes of elderly and very old critically ill patients.

We are designing a study to characterize older adults admitted to the intensive care unit and determine factors associated with adverse outcomes. The discharge registry of the ICU of a third-level hospital was reviewed. Records from January to December 2024 were reviewed. Three age groups were selected for comparison: A. <65 years; B. 65-79 years; C. 80 years and above. The outcomes to compare will be: mortality, need for invasive mechanical ventilation, ICU length of stay, and duration of mechanical ventilation.

DETAILED DESCRIPTION:
Background: Older adults represent a significant and increasing proportion of patients admitted to the intensive care unit, as the population's life expectancy is longer. The study aims to investigate factors associated with mortality in geriatric patients receiving critical care.

Methodology: We are designing a retrospective analytical cross-sectional clinical trial. The discharge records from January to December 2024 of one of the intensive care units (ICUs) from the Orinoco region in Colombia will be reviewed. The records will be divided into three groups for comparison: A. Lower than 65 years; B. between 65 and 79 years; C. 80 years and older. The records of patients admitted to the intermediate unit will be excluded. Outcomes to be evaluated will include mortality, ICU length of stay, invasive mechanical ventilation (IMV), and duration of IMV. The data will be exported to Excel. The frequency and proportion of categorical variables will be described. The central distribution and dispersion of quantitative variables will also be defined. Chi-square and Mann-Whitney U tests will be used for the statistical comparison of the variables. A value <0.05 of p will be designated as statistical significance.

Results: The frequency of older adults admitted to the ICU will be revealed at the end of the study. The outcomes and factors associated with mortality by age groups will be discriminated.

Conclusions: The study is feasible, pertinent, affordable, and essential for the region, as it will optimize resource planning and improve healthcare for critically ill older adults.

ELIGIBILITY:
Inclusion Criteria:

* Registry of adults older than 18 years, discharged from the critical care unit.

Exclusion Criteria:

* None.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults discharged from the intensive care unit during the study period, especially older adults and octogenarians.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 30 days
  Mortality during ICU stay.

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  Duration of stay in the intensive care unit
Invasive mechanical ventilation | 30 days
  Need of mechanical ventilation
Duration of IMV | 30 days
  Duration of the invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Hospital Departamental de Villavicencio
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heppner HJ, Haitham H. Intensive care of geriatric patients-a thin line between under- and overtreatment. Wien Med Wochenschr. 2022 Apr;172(5-6):102-108. doi: 10.1007/s10354-021-00902-1. Epub 2022 Jan 10. PMID 35006520
- [Result] Ball IM, Bagshaw SM, Burns KE, Cook DJ, Day AG, Dodek PM, Kutsogiannis DJ, Mehta S, Muscedere JG, Turgeon AF, Stelfox HT, Wells GA, Stiell IG. Outcomes of elderly critically ill medical and surgical patients: a multicentre cohort study. Can J Anaesth. 2017 Mar;64(3):260-269. doi: 10.1007/s12630-016-0798-4. Epub 2016 Dec 27. PMID 28028673
- [Result] Beil M, Flaatten H, Guidet B, Sviri S, Jung C, de Lange D, Leaver S, Fjolner J, Szczeklik W, van Heerden PV. The management of multi-morbidity in elderly patients: Ready yet for precision medicine in intensive care? Crit Care. 2021 Sep 10;25(1):330. doi: 10.1186/s13054-021-03750-y. PMID 34507597
- [Result] Beil M, Sviri S, Flaatten H, De Lange DW, Jung C, Szczeklik W, Leaver S, Rhodes A, Guidet B, van Heerden PV. On predictions in critical care: The individual prognostication fallacy in elderly patients. J Crit Care. 2021 Feb;61:34-38. doi: 10.1016/j.jcrc.2020.10.006. Epub 2020 Oct 13. PMID 33075607
- [Result] Shum HP, Chan KC, Wong HY, Yan WW. Outcome of elderly patients who receive intensive care at a regional hospital in Hong Kong. Hong Kong Med J. 2015 Dec;21(6):490-8. doi: 10.12809/hkmj144445. Epub 2015 Sep 29. PMID 26416174
- [Result] Rai S, Brace C, Ross P, Darvall J, Haines K, Mitchell I, van Haren F, Pilcher D. Characteristics and Outcomes of Very Elderly Patients Admitted to Intensive Care: A Retrospective Multicenter Cohort Analysis. Crit Care Med. 2023 Oct 1;51(10):1328-1338. doi: 10.1097/CCM.0000000000005943. Epub 2023 May 23. PMID 37219961
- [Result] Vincent JL, Creteur J. Appropriate care for the elderly in the ICU. J Intern Med. 2022 Apr;291(4):458-468. doi: 10.1111/joim.13371. Epub 2021 Oct 5. PMID 34487587
- [Result] Andersen FH, Ariansen Haaland O, Klepstad P, Flaatten H. Frailty and survival in elderly intensive care patients in Norway. Acta Anaesthesiol Scand. 2021 Sep;65(8):1065-1072. doi: 10.1111/aas.13836. Epub 2021 May 7. PMID 33896003
- [Result] Ramos JGR, Ranzani OT, Perondi B, Dias RD, Jones D, Carvalho CRR, Velasco IT, Forte DN. A decision-aid tool for ICU admission triage is associated with a reduction in potentially inappropriate intensive care unit admissions. J Crit Care. 2019 Jun;51:77-83. doi: 10.1016/j.jcrc.2019.02.002. Epub 2019 Feb 4. PMID 30769294
- [Result] Kim J, Choi SM, Park YS, Lee CH, Lee SM, Yim JJ, Yoo CG, Kim YW, Han SK, Lee J. Factors influencing the initiation of intensive care in elderly patients and their families: A retrospective cohort study. Palliat Med. 2016 Sep;30(8):789-99. doi: 10.1177/0269216316634241. Epub 2016 Mar 2. PMID 26934945
- [Result] Haas LEM, van Beusekom I, van Dijk D, Hamaker ME, Bakhshi-Raiez F, de Lange DW, de Keizer NF. Healthcare-related costs in very elderly intensive care patients. Intensive Care Med. 2018 Nov;44(11):1896-1903. doi: 10.1007/s00134-018-5381-8. Epub 2018 Sep 25. PMID 30255319
- [Result] Ferretti-Rebustini REL, Bispo NDS, Alves WDS, Dias TN, Santoro CM, Padilha KG. Level of acuity, severity and intensity of care of adults and older adults admitted to the Intensive Care Unit. Rev Esc Enferm USP. 2019 Jan 21;53:e03416. doi: 10.1590/S1980-220X2017051403416. English, Portuguese. PMID 30673049